CLINICAL TRIAL: NCT00664833
Title: An Open-label, Multi-center, Factorial Design, Cluster-randomized Clinical Study of Vardenafil in Canadian Males With Erectile Dysfunction: Impact of Education of the Primary Care Physician and Patient on Patient Outcomes.
Brief Title: Evaluation of LEVITRA to Advance the Treatment of Erectile Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Medical Affairs Therapeutic Area Head, Bayer HealthCare Pharmaceuticals Inc.
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: 100537; ELATED
Record Dates: First submitted 2008-04-18; First posted 2008-04-23 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Erectile Dysfunction
Keywords: Erectile dysfunction; Phosphodiesterase Type 5 Inhibitors; Patient education; Impotence; Vardenafil
MeSH Terms: conditions — Erectile Dysfunction | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 2 (Experimental)
  Interventions: Behavioral: Levitra (Vardenafil, BAY38-9456)
- Arm 4 (Other)
  Interventions: Other: No Education
- Arm 3 (Experimental)
  Interventions: Behavioral: Levitra (Vardenafil, BAY38-9456)
- Arm 1 (Experimental)
  Interventions: Behavioral: Levitra (Vardenafil, BAY38-9456)

INTERVENTIONS:
Behavioral: Levitra (Vardenafil, BAY38-9456) — The Primary Care Physician (PCP) received the educational intervention
  Arms: Arm 1
Behavioral: Levitra (Vardenafil, BAY38-9456) — The Subject received the educational intervention
  Arms: Arm 2
Behavioral: Levitra (Vardenafil, BAY38-9456) — Both the Primary Care Physician (PCP) and the subject received the educational intervention
  Arms: Arm 3
Other: No Education — No education provided to either the Primary Care Physician (PCP) or the subject.
  Arms: Arm 4

SUMMARY:
This is a multicentre, cluster-randomized, open-label flexible dose study with a 2x2 factorial design with administration of vardenafil at a dose of 5, 10 and 20 mg doses in males with erectile dysfunction.The treatment period is for 12 weeks, after a 4 week unmedicated period for subjects taking ED medication. For ED treatment-naïve subjects (ie, previously not treated with ED medication), the unmedicated period can be only 2 weeks.Approximately 150 investigational centres may be utilised with approximately 10 subjects screened and entered into a 4 week treatment free period at Visit 1 to subsequently enroll approximately 1380 subjects to therapy. Each centre should enroll 10 subjects. Sites should try to recruit approximately 50% of subjects who have not previously tried oral PDE5 inhibitor therapy for erectile dysfunction. An attempt should be made to enroll subjects whose partners are interested in being involved.Sites will be randomized in a 1:1:1:1 ratio to receive either the education intervention at the Primary care Physician (PCP) level, at the subject level, both levels or no intervention (usual care). The PCP education program is an accredited CME program and included a comprehensive overview on the screening and diagnosis of ED, the available treatment options and appropriate treatment selection, as well as subject and partner counseling. The subject education was a two-pronged approach which included physician-to-subject instruction and a direct-to-subject education method. After the unmedicated period, treatment was initiated with vardenafil 10 mg tablets for 4 weeks. This will be followed by a flexible dose titration period of 4 weeks during which subjects may maintain the previous dosage regimen or will step up to 20 mg of vardenafil or will step down to 5 mg vardenafil. There is a final 4 week treatment period where the previous dosage regimen is either maintained, increased or decreased by one step according to the three applicable dosage strengths of vardenafil (5, 10 or 20 mg). The highest applicable dosage regimen of 20 mg vardenafil will not be exceeded. A 24 hour follow-up phone call is required within 24 hours of the last dose of vardenafil to collect data concerning serious adverse events, if needed.

ELIGIBILITY:
Inclusion Criteria:

* Males with erectile dysfunction for more than six months according to the NIH Consensus Statement (the inability to attain and/or maintain penile erection sufficient for satisfactory sexual performance).
* Heterosexual relationship
* The subject must make at least four attempts at sexual intercourse (according to the question in the subject diary: "Was sexual activity initiated with the intention of intercourse?") on four separate days during the untreated baseline period.
* At least 50% of attempts during this period must be unsuccessful, according to the following questions from the subject diary [at least one question should be answered "No"]: "Were you able to achieve at least some erection (some enlargement of the penis)?", "Were you able to insert your penis into your partner's vagina?" and "Did your erection last long enough for you to have successful intercourse?"

Exclusion Criteria:

* Previous or Current Medical Conditions:

  * Any unstable medical, psychiatric or substance abuse disorder that, in the opinion of the Investigator, is likely to affect the subject's ability to complete the study or precludes the subject's participation in the study.
  * Presence of penile anatomical abnormalities (eg. penile fibrosis or Peyronie's disease) that in the opinion of the Investigator would significantly impair sexual performance.
  * History of surgical prostatectomy (transurethral interventions not excluded).
  * Hereditary degenerative retinal disorders such as retinitis pigmentosa.
  * Any underlying cardiovascular condition including unstable angina pectoris, that would preclude sexual activity.
  * Patients 65 years and older for whom the starting dose of 10 mg is judged by the investigator to be unsuitable.
  * Uncontrolled atrial fibrillation/flutter at screening (ventricular response rate of > 100 bpm).
  * Severe chronic or acute liver disease, history of moderate or severe hepatic impairment.
  * Resting hypotension (a resting systolic blood pressure of <90 mm Hg) or hypertension (a resting systolic blood pressure >170 mm Hg or a resting diastolic blood pressure >110 mm Hg).
  * Symptomatic postural hypotension within six months of Visit 1.
  * NYHA Class III or IV heart failure
* Concomitant Medications:

  * Subjects who are taking nitrates or nitric oxide donors.
  * Subjects who are taking anticoagulants, except for antiplatelet agents.
  * Subjects who are taking androgens.
  * Subjects who are taking the following inhibitors of cytochrome P 450 CYP 3A4: very potent HIV protease inhibitors (ritonavir, indinavir), the anti-mycotic agents itraconazole and ketoconazole (topical forms are allowed) or erythromycin.
  * Subjects who have received any investigational drug (including placebo) within 30 days of Visit 1.
  * Use of any treatment for erectile dysfunction within the 7 days of Visit 1 or during the study, including oral medications, vacuum devices, constrictive devices, injections or urethral suppositories.
  * Known hypersensitivity to Vardenafil, Bay 38-9456 or any component of the investigational medication.
  * Patients with a history of unresponsiveness to other PDE V inhibitor treatments due to lack of efficacy or significant side effects leading to discontinuation of the other PDE V inhibitor.
  * Subjects who are taking alpha blockers.
* Other Exclusions:

  * Subjects unwilling to cease use of vacuum devices, intracavernosal injection, Viagra or other therapy for erectile dysfunction.
  * Subjects who are unwilling or unable to complete the subject diary.
  * Subjects who are illiterate or unable to understand the questionnaires or subject diary.
  * Subjects unwilling to refrain from consuming grapefruit juice or products containing grapefruit juice with the study medication.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1029 (Actual)
Dates: Start 2004-05; Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Effect of education of the primary care physician or of the subject, in treating erectile dysfunction with vardenafil, relative to usual care, on the subject's treatment outcome of ED and quality of life. | 12 weeks

SECONDARY OUTCOMES:
To assess the safety and efficacy of vardenafil in Canadian men, when it is prescribed by the PCP, rather than specialist, and to compare the efficacy in these subgroups of subjects. | 12 weeks
To assess the effectiveness of the physician education program(s) by means of a questionnaire. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer